CLINICAL TRIAL: NCT06191731
Title: Kinetics of Urinary Excretion of Gadolinium Contrast Agents Used in MRI Examinations
Acronym: GADODURABLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Collaborators: University of Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-02-CHRMT
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Magnetic Resonance Imaging
Keywords: Contrast agents; Gadolinium; Recycling; MRI; Gadoteric acid

STUDY DESIGN:
Intervention Model Description: A single-center cohort descriptive study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- excretion kinetics of gadolinium contrast agents in patients (Experimental): urine samples are collected before Gd-CAs injection, and between 0- and two-and-a-half-hour post-injection of Gd-CAs.
  Interventions: Other: biological samples collection

INTERVENTIONS:
Other: biological samples collection — Urine samples are collected before Gd-CAs injection, and between 0- and two-and-a-half-hour post-injection of Gd-CAs.

SUMMARY:
This is a single-center cohort study aimed to describe the urinary excretion kinetics of gadolinium contrast agents (Gd-CAs). Patients with a prescription for injected MRI are invited to participate in the study. If they agree, blood and urine samples are collected before Gd-CAs injection, and urine samples are collected between 0- and two-and-a-half-hours post-injection of Gd-CAs.

DETAILED DESCRIPTION:
The contrast agents used in MRI to characterize certain lesions contain a chemical element from the rare earth family: Gadolinium (Gd). Gd, in its isolated form, is toxic in humans, but it can still be used in the form of complex molecules such as gadolinium contrast agents (Gd-CAs), which retain its contrast power while greatly minimizing its toxicity.

The MRI is performed rapidly after the injection of Gd-CAs, and these compounds are eliminated by the urinary route in the first urine following the examination. After elimination, and in view of their very high stability, these compounds follow the path of wastewater via sewage treatment plants. However, the processes currently used in these plants do not retain them, and they remain present in the purified water discharged into rivers.

Work carried out at the Laboratoire Interdisciplinaire des Environnements Continentaux (LIEC) at the University of Lorraine has demonstrated the bioaccumulation of these compounds in freshwater organisms. Gd-CAs then follow the classic pathway of continental waters. It should be noted that the quantity of Gd released as a result of MRI activities has been estimated on average at 1 injection per 1 g of Gd used.

In order to prevent future environmental disorders, recovery of all or part of the Gd-CAs immediately after MRI by urine collection is undoubtedly the most effective approach.

The aim of this project is to assess the feasibility of such an approach, and to propose a protocol applicable to MRI involving the injection of gadolinium contrast agents for urine collection.

This project is part of the "Rare Earths" theme of LabEx R21. It will examine the possibility of recycling gadolinium as an element or as Gd-CAs.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* over 18 years of age
* with a prescription for MRI with gadolinium-based contrast agents (Gd-CAs) injection validated by a radiologist
* affiliated with a health insurance plan
* have signed an informed consent form

Exclusion Criteria:

* Patients:
* with known allergy to gadolinium-based contrast agents (Gd-CAs)
* with known severe renal impairment (GFR < 30 mL/min)
* on dialysis
* with urinary incontinence
* with an ongoing urinary tract infection
* under hydric or hydrosodic restriction
* unable to urinate independently
* Protected persons (under guardianship, curatorship or safeguard of justice)
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-04-12 (Estimated); Study Completion 2026-04-12 (Estimated)

PRIMARY OUTCOMES:
Urinary excretion of gadolinium-based contrast agents (Gd-CAs) | at 2 hours and a half after Gd-CAs injection
  Describe the kinetics of urinary excretion of GdCAs during the 2H30 following gadoline contrast injection in patients undergoing injected MRI at the Mercy Hospital Medical Imaging Department.
  The cumulative quantity of gadolinium-based contrast agents (Gd-CAs) (mg) mesured in urine during spontaneous micturition between 0 and 2H30 after injection of gadoline contrast medium and during micturition on demand at 2.30 h. The amount of Gd present in the urine (directly associated with the presence of Gd-CAs) is determined by inductively coupled plasma mass spectrometry (ICPMS). Urine concentrations are expressed in µg/L. Taking into account the volume of urine collected, the quantity of Gd is calculated and expressed in mg. This quantity is then expressed as a percentage of the quantity of injected-Gd-CAs.

SECONDARY OUTCOMES:
Renal function | Day 0 (MRI)
  Glomerular filtration rate (GFR: mL/min) estimated by the CKD-EPI method on the day of MRI.
Volume of beverages | at 2 hours and a half after Gd-CAs injection
  Volume of beverages drunk (mL) after each micturition, declared by the patient since Gd-CAs injection, to the nearest 100 mL.
Time to first spontaneous micturition | up to 2 hours and a half after Gd-CAs injection
  Duration (in minutes) between time of Gd-CAs injection and time of first spontaneous micturition.
Study refusal rate | Day 0 (MRI)
  Percentage (%) of study refusal
Rate of premature study exit | at 2 hours and a half after Gd-CAs injection
  Percentage (%) of premature study exit

CONTACTS AND LOCATIONS:
Overall Officials: Rémi DUPRES, MD, Principal Investigator — CHR Metz Thionville Hopital Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, Grand Est, France

IPD SHARING:
Plan to Share IPD: No